CLINICAL TRIAL: NCT04247971
Title: Pulmonary Inflammation and Microbiome Changes With Bariatric Surgery in Obese Asthma
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00104326
Record Dates: First submitted 2020-01-27; First posted 2020-01-30 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Asthma; Obesity
MeSH Terms: conditions — Asthma; Obesity | interventions — Blood Specimen Collection; Respiratory Physiological Phenomena

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and sputum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Obese, early-onset asthmatics: Obese adults (BMI>or= 30) between the ages of 21-60 with an initial asthma diagnosis at <12 years of age
  Interventions: Procedure: Blood draw; Procedure: Sputum collection; Procedure: Pulmonary function test
- Obese, late-onset asthmatics: Obese adults (BMI > or = 30) between the ages of 21-60 with an initial asthma diagnosis at >12 years of age
  Interventions: Procedure: Blood draw; Procedure: Sputum collection; Procedure: Pulmonary function test
- Obese non-asthmatics: Obese adults (BMI > or = 30) between the ages of 21-60 with no asthma diagnosis
  Interventions: Procedure: Blood draw; Procedure: Sputum collection; Procedure: Pulmonary function test

INTERVENTIONS:
Procedure: Blood draw — 23 ml of blood collected
Procedure: Sputum collection — Induced sputum sample collected
Procedure: Pulmonary function test — Pulmonary function testing

SUMMARY:
The purpose of this study is to gain understanding of mechanisms whereby bariatric surgery modulates pulmonary inflammation and pulmonary microbiome composition and how these changes direct the pathobiology of human obese asthma.

ELIGIBILITY:
Inclusion Criteria:

Asthma Subjects

* Outpatient adults of either sex 21-60 years of age with an initial asthma diagnosis at < 12 years of age (early-onset) or >12 years of age (late-onset), as defined by the NHLBI NAEPP guidelines (17).
* Subjects with obesity (BMI ≥ 30 kg/m2).
* Physician diagnosis of asthma.
* Eligible and scheduled for bariatric surgery (Roux-en-Y gastric bypass, sleeve gastrectomy or duodenal switch) and receiving care within the Duke Health System.

FEV1 within acceptable limits (>45% predicted before and >55% predicted after, bronchodilator administration).

* Relatively healthy subjects able to undergo sputum induction without complications.
* Willing and able to give informed consent and adhere to visit/protocol schedules.
* Read and write in English.

Non-Asthma Control Subjects

* Outpatient adults of either sex 21-60 years of age.
* Subjects with obesity (BMI ≥ 30).
* Eligible and scheduled for bariatric surgery (Roux-en-Y gastric bypass, sleeve gastrectomy or duodenal switch) at Duke Regional Hospital and receiving care at the Duke Metabolic and -Weight Loss Surgery Center.
* Normal lung function.
* No clinical history of atopy.
* No significant medical or psychological issues.
* Healthy subjects able to undergo sputum induction without complications.
* Willing and able to give informed consent and adhere to visit/protocol schedules.
* Read and write in English.

Exclusion Criteria:

* Children < 21 years of age.
* Inpatient status.
* Ineligibility or not scheduled for bariatric surgery at the Duke Metabolic and Weight Loss Surgery Center.
* FEV1 is less than 45% predicted before, or less than 55% predicted after, bronchodilator administration.
* Upper or lower respiratory tract infection within one month of the study.
* Use of systemic corticosteroids within four weeks of study.
* Smoking (tobacco, e-cigarette, vaping or inhaled drugs) history > 5 pack years or smoking or vaping within the previous six months.
* Significant non-asthma pulmonary disease (stable obstructive sleep apnea is not excluded).
* An ED visit or inpatient admission for a primary respiratory diagnosis within 60 days of enrollment.
* Poorly controlled concomitant conditions that pose additional procedure risk as determined by the investigator.
* All patients on anticoagulants.
* Uncontrolled sleep apnea.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Cohort of 15-20 obese, early-onset asthmatic, 15-20 obese, late-onset asthmatic, and 15-20 obese non-asthmatic subjects will be recruited. Subjects in each group will undergo an initial screening visit (V0) to establish the subject groups according to asthma diagnosis, asthma onset age and type of scheduled surgery.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2021-04-30 (Actual); Primary Completion 2023-02-09 (Actual); Study Completion 2023-02-09 (Actual)

PRIMARY OUTCOMES:
Change in leptin levels | Baseline (2 weeks before surgery), 30 days post-surgery, 3 months post-surgery
Change in adiponectin levels | Baseline (2 weeks before surgery), 30 days post-surgery, 3 months post-surgery
Change in IL-8 levels | Baseline (2 weeks before surgery), 30 days post-surgery, 3 months post-surgery
Change in IL-6 levels | Baseline (2 weeks before surgery), 30 days post-surgery, 3 months post-surgery
Change in cystatin-c levels | Baseline (2 weeks before surgery), 30 days post-surgery, 3 months post-surgery
Change in IL-17 levels | Baseline (2 weeks before surgery), 30 days post-surgery, 3 months post-surgery
Change in IL-1beta levels | Baseline (2 weeks before surgery), 30 days post-surgery, 3 months post-surgery
Change in TNF-α levels | Baseline (2 weeks before surgery), 30 days post-surgery, 3 months post-surgery
Change in YKL-40 levels | Baseline (2 weeks before surgery), 30 days post-surgery, 3 months post-surgery
Change in lung function as measured by forced expiratory volume | Baseline (2 weeks before surgery), 30 days post-surgery, 3 months post-surgery
Change in lung function as measured by forced vital capacity | Baseline (2 weeks before surgery), 30 days post-surgery, 3 months post-surgery
Change in lung function as measured by fractional concentration of exhaled nitro oxide | Baseline (2 weeks before surgery), 30 days post-surgery, 3 months post-surgery
Change in lung function as measured by FEV1/FVC | Baseline (2 weeks before surgery), 30 days post-surgery, 3 months post-surgery
Change in lung function as measured by forced expiratory flow | Baseline (2 weeks before surgery), 30 days post-surgery, 3 months post-surgery

CONTACTS AND LOCATIONS:
Overall Officials: Kunoor Jain-Spangler, MD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No